CLINICAL TRIAL: NCT01654380
Title: Comparison of the Effects of LY2605541 and Insulin Glargine on Endogenous Glucose Output and Peripheral Glucose Disposal in Healthy Subjects and Patients With Type 1 Diabetes Mellitus
Brief Title: A Study of LY2605541 Versus Insulin Glargine on Blood Sugar
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 12157; I2R-MC-BIAV (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Results first posted 2019-03-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2018-11

CONDITIONS: Healthy Volunteers; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — LY2605541; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part A, Cohort A; LY2605541 (Experimental): Healthy participants received 5.1 milliunits/minute (mU/min) in Period 1, 10.2 mU/min in Period 2, and 15.3 mU/min in Period 3, administered intravenously (IV) over 8 hours. All periods were separated by a minimum 6-day washout period
  Interventions: Drug: LY2605541
- Part A, Cohort A; Insulin Glargine (Active Comparator): Healthy participants received insulin glargine (30 milliunits/meter squared/minute [mU/m^2/min]) administered IV over 8 hours in Period 4. All periods were separated by a minimum 6-day washout period
  Interventions: Other: Insulin glargine
- Part A, Cohort B; LY2605541 (Experimental): Healthy participants received 15.3 mU/min in Period 1, 37.0 mU/min in Period 2, and 74.1 mU/min in Period 3, administered IV over 8 hours. All periods were separated by a minimum 6-day washout period.
  Interventions: Drug: LY2605541
- Part A, Cohort B; Insulin Glargine (Active Comparator): Healthy participants received insulin glargine (60 mU/m^2/min) administered IV over 8 hours in Period 4. All periods were separated by a minimum 6-day washout period.
  Interventions: Other: Insulin glargine
- Part B; LY2605541 (Experimental): Participants with T1DM received 15.3 mU/min in 1 of 4 study periods, administered IV up to 8 hours and received 74.1 mU/min in 1 of 4 Periods, administered IV up to 10 hours. Each dose was separated by a minimum 6-day washout period.
  Interventions: Drug: LY2605541
- Part B; Insulin Glargine (Active Comparator): Participants with T1DM received 1 insulin glargine dose per study period (10 and 20 mU/m^2/min) administered IV over 8 hours in 2 of 4 study periods. Each dose was separated by a minimum 6-day washout period.
  Interventions: Other: Insulin glargine

INTERVENTIONS:
Drug: LY2605541 — LY2605541 is a solution. The concentration of LY2605541 is 100 units/milliliter (U/mL).
  Arms: Part A, Cohort A; LY2605541; Part A, Cohort B; LY2605541; Part B; LY2605541
Other: Insulin glargine — Insulin glargine is a 100 U/mL solution in 10 milliliter (mL) glass vial.
  Arms: Part A, Cohort A; Insulin Glargine; Part A, Cohort B; Insulin Glargine; Part B; Insulin Glargine

SUMMARY:
LY2605541 is an investigational drug being developed for the treatment of diabetes mellitus. This study is designed to understand how the body handles the investigational drug, what effect this investigational drug has on the body, and how much should be given. This study will also measure how much of the investigational drug gets into the blood stream and how long it takes the body to get rid of it. The study has 2 parts: Part A will be conducted in healthy participants. Part B will be conducted in participants with type 1 diabetes mellitus (T1DM). This study will take approximately 10-14 days spread over 6-20 weeks, not including screening. Screening will be performed within 30 days of the start of the study.

ELIGIBILITY:
Inclusion Criteria:

All Participants

* Are healthy males or participants with T1DM
* Have a screening body mass index (BMI) of 20.0-29.9 kilograms per square meter (kg/m^2)

Healthy Participants ONLY

* Are overtly healthy, as determined by medical history and physical examination
* Have a fasting blood glucose <108 milligrams/deciliter (mg/dL) (6.0 millimoles/liter [mmol/L]) at screening

Participants with T1DM ONLY

* Have a diagnosis of T1DM for at least 1 year based on medical history
* Have a screening c-peptide <0.5 nanograms/milliliter (ng/mL)
* Have a hemoglobin A1c (HbA1c) of 6.0 to 9.0% at screening
* Have had no episodes of severe hypoglycemia in the past 6 months

Exclusion Criteria:

All Participants

* Have a hemoglobin level <12.0 grams/deciliter (g/dL)
* Are currently a smoker, used tobacco products on a regular basis in the 6 months prior to screening, or are intending to smoke during the study

Healthy Participants ONLY

• Regular use or intended use of over-the counter or prescription medication within 7 and 14 days, respectively, prior to dosing (apart from vitamin/mineral supplements or occasional use of acetaminophen or ibuprofen).

Participants with T1DM ONLY

* Regular use or intended use of any over-the-counter or prescription medications or nutritional supplements that affect blood glucose or the body's sensitivity to insulin or that promote weight loss within 14 days prior to dosing
* Are receiving chronic (lasting longer than 14 consecutive days) systemic or inhaled glucocorticoid therapy (excluding topical, intra-articular, and intraocular preparations) or have received such therapy within the 4 weeks before dosing
* Require a total daily insulin dose exceeding 100 units (U)
* Have fasting triglycerides >400 mg/dL

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A, Cohort A: LY2605541 First, Then Insulin Glargine: LY2605541: Healthy participants received 5.1 milliunits/minute (mU/min) in Period 1, 10.2 mU/min in Period 2, and 15.3 mU/min in Period 3, administered intravenously (IV) over 8 hours.
  Insulin glargine: Healthy participants received 30 milliunits/meter squared/minute [mU/m^2/min]) administered IV over 8 hours in Period 4
- Part A, Cohort B: LY2605541 First, Then Insulin Glargine: LY2605541: Healthy participants received 15.3 mU/min in Period 1, 37.0 mU/min in Period 2, and 74.1 mU/min in Period 3, administered IV over 8 hours.
  Insulin glargine: Healthy participants received 20 mU/m^2/min administered IV over 8 hours in Period 4
- Part B: LY2605541: LY2605541: Participants with T1DM received 15.3 mU/min in 1 of 4 Periods, administered IV up to 8 hours and received 74.1 mU/min in 1 of 4 Periods, administered IV up to 10 hours.
- Part B: Insulin Glargine: Insulin glargine: Participants with T1DM received 10 mU/m^2/min in 1 of 4 Periods and received 20 mU/m^2/min in 1 of 4 Periods, administered IV over 8 hours.
Period: Part A, Period 1
Arm/Group | Part A, Cohort A: LY2605541 First, Then Insulin Glargine | Part A, Cohort B: LY2605541 First, Then Insulin Glargine | Part B: LY2605541 | Part B: Insulin Glargine
Started | 4 | 4 | 0 | 0
Received at Least 1 Dose of Study Drug | 4 | 4 | 0 | 0
Completed | 4 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part A, Washout of at Least 6 Days
Arm/Group | Part A, Cohort A: LY2605541 First, Then Insulin Glargine | Part A, Cohort B: LY2605541 First, Then Insulin Glargine | Part B: LY2605541 | Part B: Insulin Glargine
Started | 4 | 4 | 0 | 0
Completed | 4 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part A, Period 2
Arm/Group | Part A, Cohort A: LY2605541 First, Then Insulin Glargine | Part A, Cohort B: LY2605541 First, Then Insulin Glargine | Part B: LY2605541 | Part B: Insulin Glargine
Started | 4 | 4 | 0 | 0
Completed | 4 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part A, Washout of at Least 6 Days
Arm/Group | Part A, Cohort A: LY2605541 First, Then Insulin Glargine | Part A, Cohort B: LY2605541 First, Then Insulin Glargine | Part B: LY2605541 | Part B: Insulin Glargine
Started | 4 | 4 | 0 | 0
Completed | 4 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part A, Period 3
Arm/Group | Part A, Cohort A: LY2605541 First, Then Insulin Glargine | Part A, Cohort B: LY2605541 First, Then Insulin Glargine | Part B: LY2605541 | Part B: Insulin Glargine
Started | 4 | 4 | 0 | 0
Completed | 4 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part A, Washout of at Least 6 Days
Arm/Group | Part A, Cohort A: LY2605541 First, Then Insulin Glargine | Part A, Cohort B: LY2605541 First, Then Insulin Glargine | Part B: LY2605541 | Part B: Insulin Glargine
Started | 4 | 4 | 0 | 0
Completed | 4 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part A, Period 4
Arm/Group | Part A, Cohort A: LY2605541 First, Then Insulin Glargine | Part A, Cohort B: LY2605541 First, Then Insulin Glargine | Part B: LY2605541 | Part B: Insulin Glargine
Started | 4 | 4 | 0 | 0
Completed | 4 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part B, Period 1
Arm/Group | Part A, Cohort A: LY2605541 First, Then Insulin Glargine | Part A, Cohort B: LY2605541 First, Then Insulin Glargine | Part B: LY2605541 | Part B: Insulin Glargine
Started | 0 (Participants in Part A were not included in Part B.) | 0 (Participants in Part A were not included in Part B.) | 7 (Participants in Part B were not included in Part A.) | 7 (Participants in Part B were not included in Part A.)
Received at Least 1 Dose of Study Drug | 0 | 0 | 7 | 7
Completed | 0 | 0 | 6 (Participant who did not complete received only 1 dose of LY2605541 74.1 mU/min IV for 8 hours) | 7
Not Completed | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Period: Part B, Washout of at Least 6 Days
Arm/Group | Part A, Cohort A: LY2605541 First, Then Insulin Glargine | Part A, Cohort B: LY2605541 First, Then Insulin Glargine | Part B: LY2605541 | Part B: Insulin Glargine
Started | 0 | 0 | 6 | 7
Completed | 0 | 0 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Part B, Period 2
Arm/Group | Part A, Cohort A: LY2605541 First, Then Insulin Glargine | Part A, Cohort B: LY2605541 First, Then Insulin Glargine | Part B: LY2605541 | Part B: Insulin Glargine
Started | 0 | 0 | 6 | 7
Completed | 0 | 0 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Part B, Washout of at Least 6 Days
Arm/Group | Part A, Cohort A: LY2605541 First, Then Insulin Glargine | Part A, Cohort B: LY2605541 First, Then Insulin Glargine | Part B: LY2605541 | Part B: Insulin Glargine
Started | 0 | 0 | 6 | 7
Completed | 0 | 0 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Part B, Period 3
Arm/Group | Part A, Cohort A: LY2605541 First, Then Insulin Glargine | Part A, Cohort B: LY2605541 First, Then Insulin Glargine | Part B: LY2605541 | Part B: Insulin Glargine
Started | 0 | 0 | 6 | 7
Completed | 0 | 0 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Part B, Washout of at Least 6 Days
Arm/Group | Part A, Cohort A: LY2605541 First, Then Insulin Glargine | Part A, Cohort B: LY2605541 First, Then Insulin Glargine | Part B: LY2605541 | Part B: Insulin Glargine
Started | 0 | 0 | 6 | 7
Completed | 0 | 0 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Part B, Period 4
Arm/Group | Part A, Cohort A: LY2605541 First, Then Insulin Glargine | Part A, Cohort B: LY2605541 First, Then Insulin Glargine | Part B: LY2605541 | Part B: Insulin Glargine
Started | 0 | 0 | 6 | 7
Completed | 0 | 0 | 6 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A: All participants who received at least 1 dose of study drug in Part A of the study.
- Part B: All participants who received at least 1 dose of study drug in Part B of the study.
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Total
Number analyzed (Participants) | 8 | 14 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (1.5) | 34.7 (10.5) | 31.6 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 14 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  White | 7 | 14 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 14 | 22

OUTCOME MEASURES:

1. Primary Outcome: Part B: Glucodynamics: Endogenous Glucose Output
Description: The percent suppression from baseline in endogenous glucose production (EGP) is presented. Percent EGP change from baseline was calculated by (1-[last 2 hours of EGP/basal EGP])*100.
  The duration of the clamp procedure was 10 hours for the LY2605541 74.1 mU/min dose in Part B. The duration of the clamp procedures performed at the 15.3 mU/min LY2605541 dose and both of the insulin glargine doses was 8 hours.
Time Frame: Baseline, up to 10 hours (duration of the euglycemic glucose clamp)
Population: Participants who received at least 1 dose of study drug with evaluable EGP data
Measure: Mean (Standard Deviation); unit: percent of suppression
Groups:
- 15.3 mU/Min LY2605541: LY2605541: Participants with T1DM received 15.3 mU/min in 1 of 4 Periods in Part B, administered IV for up to 8 hours
- 74.1 mU/Min LY2605541: LY2605541: Participants with T1DM received 74.1 mU/min in 1 of 4 Periods in Part B, administered IV for up to 10 hours
- 10 mU/m^2/Min Insulin Glargine: Insulin glargine: Participants with T1DM received 10 mU/m^2/min in 1 of 4 Periods in Part B, administered IV over 8 hours
- 20 mU/m^2/Min Insulin Glargine: Insulin glargine: Participants with T1DM received 20 mU/m^2/min in 1 of 4 Periods in Part B, administered IV over 8 hours
Arm/Group | 15.3 mU/Min LY2605541 | 74.1 mU/Min LY2605541 | 10 mU/m^2/Min Insulin Glargine | 20 mU/m^2/Min Insulin Glargine
Number analyzed (Participants) | 14 | 13 | 13 | 12
percent of suppression | 64.53 (19.35) | 99.23 (1.76) | 78.05 (17.33) | 97.05 (6.47)

2. Primary Outcome: Part B: Glycodynamics: Glucose Disposal
Description: The fold change from baseline in glucose disappearance rate (GDR) is presented. The fold GDR increase from baseline was calculated by last 2 hours of GDR/basal GDR.
  The duration of the clamp procedure was 10 hours for the LY2605541 74.1 mU/min dose in Part B. The duration of the clamp procedures performed at the 15.3 mU/min LY2605541 dose and both of the insulin glargine doses was 8 hours.
Time Frame: Baseline, up to 10 hours (duration of the euglycemic glucose clamp)
Population: Participants who received at least 1 dose of study drug with evaluable GDR data.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | 15.3 mU/Min LY2605541 | 74.1 mU/Min LY2605541 | 10 mU/m^2/Min Insulin Glargine | 20 mU/m^2/Min Insulin Glargine
Number analyzed (Participants) | 14 | 13 | 13 | 12
fold change | 0.68 (0.09) | 1.42 (0.35) | 0.98 (0.39) | 1.85 (0.59)

3. Primary Outcome: Part B: Glycodynamics: Maximum Rate of Glucose Disposal
Description: The maximum rate of glucose disposal (Rdmax) is presented. The duration of the clamp procedure was 10 hours for the LY2605541 74.1 mU/min dose in Part B. The duration of the clamp procedures performed at the 15.3 mU/min LY2605541 dose and both of the insulin glargine doses was 8 hours.
Time Frame: Baseline, up to 10 hours (duration of the euglycemic glucose clamp)
Population: Participants who received at least 1 dose of study drug with evaluable Rdmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams/minute/kilograms (mg/min/kg)
Arm/Group | 15.3 mU/Min LY2605541 | 74.1 mU/Min LY2605541 | 10 mU/m^2/Min Insulin Glargine | 20 mU/m^2/Min Insulin Glargine
Number analyzed (Participants) | 14 | 13 | 13 | 13
milligrams/minute/kilograms (mg/min/kg) | 1.80 (24) | 2.89 (23) | 2.15 (28) | 3.55 (40)

ADVERSE EVENTS:
Groups:
- Part A, Cohort A: 5.1 mU/Min LY2605541: LY2605541: Healthy participants received 5.1 mU/min in Period 1, administered IV over 8 hours
- Part A, Cohort A: 10.2 mU/Min LY2605541: LY2605541: Healthy participants received 10.2 mU/min in Period 2, administered IV over 8 hours
- Part A, Cohort A or Cohort B: 15.3 mU/Min LY2605541: LY2605541: Healthy participants received 15.3 mU/min in Period 3 of Part A Cohort A and 15.3 mU/min in Period 1 of Part A Cohort B, administered IV over 8 hours
- Part A, Cohort A: 30 mU/m^2/Min Insulin Glargine: Insulin glargine: Healthy participants received 30 mU/m^2/min administered IV over 8 hours in Period 4
- Part A, Cohort B: 37.0 mU/Min LY2605541: LY2605541: Healthy participants received 37.0 mU/min in Period 2 administered IV over 8 hours
- Part A, Cohort B: 74.1 mU/Min LY2605541: LY2605541: Healthy participants received 74.1 mU/min in Period 3, administered IV over 8 hours
- Part A, Cohort B: 20 mU/m^2/Min Insulin Glargine: Insulin glargine: Healthy participants received 20 mU/m^2/min administered IV over 8 hours in Period 4
- Part B: 15.3 mU/Min LY2605541: LY2605541: Participants with T1DM received 15.3 mU/min in 1 of 4 Periods in Part B, administered IV for up to 10 hours
- Part B: 74.1 mU/Min LY2605541: LY2605541: Participants with T1DM received 74.1 mU/min in 1 of 4 Periods in Part B, administered IV for up to 10 hours
- Part B: 10 mU/m^2/Min Insulin Glargine: Insulin glargine: Participants with T1DM received 10 mU/m^2/min in 1 of 4 Periods in Part B, administered IV over 8 hours
- Part B: 20 mU/m^2/Min Insulin Glargine: Insulin glargine: Participants with T1DM received 20 mU/m^2/min in 1 of 4 Periods in Part B, administered IV over 8 hours
Arm/Group | Part A, Cohort A: 5.1 mU/Min LY2605541 | Part A, Cohort A: 10.2 mU/Min LY2605541 | Part A, Cohort A or Cohort B: 15.3 mU/Min LY2605541 | Part A, Cohort A: 30 mU/m^2/Min Insulin Glargine | Part A, Cohort B: 37.0 mU/Min LY2605541 | Part A, Cohort B: 74.1 mU/Min LY2605541 | Part A, Cohort B: 20 mU/m^2/Min Insulin Glargine | Part B: 15.3 mU/Min LY2605541 | Part B: 74.1 mU/Min LY2605541 | Part B: 10 mU/m^2/Min Insulin Glargine | Part B: 20 mU/m^2/Min Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/8 | 0/4 | 0/4 | 0/4 | 0/4 | 0/14 | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/4 | 2/4 | 3/8 | 2/4 | 1/4 | 0/4 | 1/4 | 1/14 | 3/13 | 2/13 | 5/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Cohort A: 5.1 mU/Min LY2605541 (N=4) | Part A, Cohort A: 10.2 mU/Min LY2605541 (N=4) | Part A, Cohort A or Cohort B: 15.3 mU/Min LY2605541 (N=8) | Part A, Cohort A: 30 mU/m^2/Min Insulin Glargine (N=4) | Part A, Cohort B: 37.0 mU/Min LY2605541 (N=4) | Part A, Cohort B: 74.1 mU/Min LY2605541 (N=4) | Part A, Cohort B: 20 mU/m^2/Min Insulin Glargine (N=4) | Part B: 15.3 mU/Min LY2605541 (N=14) | Part B: 74.1 mU/Min LY2605541 (N=13) | Part B: 10 mU/m^2/Min Insulin Glargine (N=13) | Part B: 20 mU/m^2/Min Insulin Glargine (N=13)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days